CLINICAL TRIAL: NCT01914445
Title: Chromoendoscopy of the Colon After Oral Administration of Indigo Carmine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HYMC-46-13
Record Dates: First submitted 2013-07-31; First posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Indigo Carmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Indigo Carmine (Experimental): Indigo Carmine (2 mg per kilo) and 2nd half of PEG dose will be orally administered to patients prior to colonoscopy.
  Interventions: Drug: Indigo Carmine

INTERVENTIONS:
Drug: Indigo Carmine — Oral administration of Indigo Carmine prior to colonoscopy
  Other Names: FD&C Blue 2

SUMMARY:
The purpose of this study is to examine whether oral administration of Indigo Carmine together with Polyethylene Glycol (PEG), the usual colon preparatory solution, can be used instead of staining during the examination itself.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Inflammatory Bowel Disease
* Patients under surveillance for Disease-Associated Lesions and Masses (DALM)

Exclusion Criteria:

* All others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Indigo Carmine during oral administration | One hour
  The efficacy of Indigo Carmine in staining tissues to better characterize, delineate, and highlight the gastrointestinal mucosa will be determined during the colonoscopic examination. Biopsies will be taken from suspicious lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Verzhbitsky, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel